CLINICAL TRIAL: NCT02731261
Title: Chronic Effects of Exercise on Motor Memory Consolidation in Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Castelo Branco (Other)
Responsible Party: Principal Investigator, André Ramalho, Mss, Instituto Politécnico de Castelo Branco
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESE IPCB01
Record Dates: First submitted 2016-03-23; First posted 2016-04-07 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Elderly

ARMS (2):
- Experimental (Experimental)
  Interventions: Other: Motor memory consolidation
- Control (No Intervention)

INTERVENTIONS:
Other: Motor memory consolidation — Subjects were divided in two groups: a control group and an experimental group. Before the intervention of a physical exercise program, subjects performed a Finger Tapping Sequence to measure baseline performance. After the intervention, the assessment of the impact of exercise on motor memory consolidation was held in three stages: Training; 1 hour after training and 24 hours after training.
  Arms: Experimental

SUMMARY:
The main purpose of this study was to investigate if a six months period of physical exercise could improve motor memory consolidation in elderly people.

DETAILED DESCRIPTION:
38 subjects of both genders, with a mean age of 71 years old participated in the study. Subjects were divided in two groups: a control group and an experimental group. Before the intervention of a physical exercise program, subjects performed a Finger Tapping Sequence to measure baseline performance. After the intervention, the assessment of the impact of exercise on motor memory consolidation was held in three stages: Training; 1 hour after training and 24 hours after training.

ELIGIBILITY:
Inclusion Criteria:

* individuals not engaged in physical activity;
* persons aged from 65 years.

Exclusion Criteria:

* sensory abnormalities;
* mental abnormalities;
* motor abnormalities;
* other atypical health problems.

Ages: 65 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Subjects performed a Finger Tapping Sequence to measure a performance in Motor memory consolidation. | 6 months
  The participants were required to learn a Finger Tapping Sequence (4_1_3_2_4) by using a computer keyboard. The finger sequence corresponded to computer keys as follows: digit 1 - Index finger; digit 2 - Middle finger; digit 3 - Ring finger; digit 4 - Little. The participants were requested to repeat the sequence as quickly and as accurately as possible for 30 seconds.